CLINICAL TRIAL: NCT04471935
Title: Speech Hero: a Rhythm-based Speech Therapy App for Individuals With Aphasia
Brief Title: Speech Hero Home Therapy for Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flint Rehabilitation Devices, LLC (Industry)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1R43DC018771-01 (NIH)
Record Dates: First submitted 2020-07-07; First posted 2020-07-15 (Actual); Results first posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Broca Aphasia
MeSH Terms: conditions — Aphasia, Broca

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- At home Speech Hero therapy (Other)
  Interventions: Device: At home Speech Hero therapy app

INTERVENTIONS:
Device: At home Speech Hero therapy app — Participants will be instructed to use the Speech Hero therapy app for three hours per week over a 4-week period.

SUMMARY:
The investigators will run an at-home usability study of a newly developed speech therapy app called Speech Hero with 10 individuals with Broca's aphasia in the chronic stage of stroke. The Speech Hero app allows users to perform rhythm-based speech exercises at home. For this study participants will be instructed to use Speech Hero for at least 10 hours over a 4-week period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Broca's aphasia due to stroke,
* >6 months post stroke
* sufficient motor function of the unaffected upper extremity to tap on a table while speaking

Exclusion Criteria:

* Incidence of other neurological diseases (though individuals with apraxia will be included)
* age <85

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yune Lee, PhD, Principal Investigator — University of Texas
Locations (1):
- Callier Center at University of Texas Dallas, Richardson, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- At Home Speech Hero Therapy: At home Speech Hero therapy app: Participants will be instructed to use the Speech Hero therapy app for three hours per week over a 3-week period.
Period: Overall Study
Arm/Group | At Home Speech Hero Therapy
Started | 10
Completed | 8
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Deemed ineligible to participate | 1

BASELINE CHARACTERISTICS:
Arm/Group | At Home Speech Hero Therapy
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Used the Device for at Least Ten Hours Over the Course of Four Weeks
Description: Number of participants able to use the device on their own at home for at least 10 hours over four weeks without technical or other issues. Speech Hero will be deemed feasible for this population if at least 5 participants are able to use the device on their own at home for at least 10 hours over four weeks without technical or other issues.
Time Frame: Immediately Post-Treatment, an average of 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- At Home Speech Hero Therapy: At home Speech Hero therapy app: Participants will be instructed to use the Speech Hero therapy app for at least 10 hours over a 4-week period.
Arm/Group | At Home Speech Hero Therapy
Number analyzed (Participants) | 8
Participants | 7

2. Secondary Outcome: Change in Score on Western Aphasia Battery
Description: Assessment of language function of adults with suspected neurological disorders as a result of a stroke, head injury, or dementia. The Western Aphasia Battery (WAB) is comprised of 8 subscales. For this study the subscales of spontaneous speech, auditory verbal comprehension, repetition, naming and word finding were used. Results reported as change in score from baseline to post-treatment (each subscale score is on 0-100% scale with higher score representing less impairment).
Time Frame: Immediately Post-Treatment, an average of 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | At Home Speech Hero Therapy
Number analyzed (Participants) | 8
score on a scale
  Spontaneous Speech | 3 (7)
  Auditory Verbal Comprehension | -1 (7)
  Repetition | 2 (10)
  Naming and Word Finding | 6 (4)

3. Secondary Outcome: Change in Score on Boston Naming Test
Description: Assessment of language function of adults with suspected neurological disorders as a result of a stroke, head injury, or dementia. Scoring counts the number of spontaneously produced correct responses, the number of cues given, and the number of responses after phonemic cueing and after semantic cueing. Results reported as change in score from baseline to post-treatment (score for Boston Naming Test (BNT) is on 0-100% scale with higher score representing less impairment).
Time Frame: Immediately Post-Treatment, an average of 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | At Home Speech Hero Therapy
Number analyzed (Participants) | 8
score on a scale | 5 (9)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | At Home Speech Hero Therapy
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT04471935/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT04471935/ICF_001.pdf